CLINICAL TRIAL: NCT01209429
Title: Importance of the GH/IGF-1 Axis for Human Substrate and Energy Metabolism During Calorie Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Birgitte Nellemann, MD PhD student, University of Aarhus
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: M-20100150
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Calorie restriction; GH/IGF-I axis; STATb5; SIRT1; Intracellular signaling peptides and proteins; Fasting; Growth hormone; IGF-1
MeSH Terms: conditions — Fasting | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 42 hour fast/GH infusion (Experimental)
  Interventions: Drug: GH hormone infusion; Behavioral: 42 hour fast
- 42 hour fast/Placebo infusion (Experimental)
  Interventions: Behavioral: 42 hour fast
- 12 hour fast/GH infusion (Experimental)
  Interventions: Drug: GH hormone infusion; Behavioral: 12 hour fast
- 12 hour fast/Placebo infusion (Placebo Comparator)
  Interventions: Behavioral: 12 hour fast

INTERVENTIONS:
Drug: GH hormone infusion — Norditropin 30 ng/kg/min
  Other Names: Norditropin; Genotropin
  Arms: 12 hour fast/GH infusion; 42 hour fast/GH infusion
Behavioral: 42 hour fast — The participant will be fasting 42 hours prior to the start of the study day, drinking water is allowed
  Other Names: No other name
  Arms: 42 hour fast/GH infusion; 42 hour fast/Placebo infusion
Behavioral: 12 hour fast — 12 hour fast will be used as a control scenario to 42 hour fast
  Other Names: No other name
  Arms: 12 hour fast/GH infusion; 12 hour fast/Placebo infusion

SUMMARY:
This study will investigate whether growth hormone is modulated by the enzyme SIRT1 and by that is stimulating lipolysis on expense of IGF-I production. This is done in 10 healthy men on calorie restriction on 4 study days with fat and skeletal muscle biopsies.

DETAILED DESCRIPTION:
It has been shown that calorie restriction enhances the length of life in yeast, worms, fish and rodent. Whether this elongation of life due to calorie restriction can be applied to humans is not known. However, it is a fact that calorie restriction will decrease the risk of developing metabolic disturbances such as diabetes, hypertension and atherosclerosis.

On the molecular level the specific relations are not fully understood. This study will investigate the possible connection between SITR1 and the relation to the GH/IGF-I axis and STAT5b in healthy men. The participant will fast 42 and 12 hours respectively, and have GH or placebo infusions. The design is a classical 2x2 design and will be randomized.

Knowledge of the interactions between calorie restriction, SIRT1, STAT5b and the GH/IGF-I axis will apply important information about the relations between aging, energy metabolism and metabolic disturbances.

ELIGIBILITY:
Inclusion Criteria:

* healthy lean men
* age >18

Exclusion Criteria:

* metabolic disturbances
* alcohol drug abuse
* malign disease: current or previous

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Description of intracellular pathways to clarify the interplay between calorie restriction, SIRT1, STATb5, and the GH/IGF-I axis | 6 hour study days
  All study days consists of 3 hour basic periods and 3 hours hyperinsulinemic, euglycemic clamp.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Professor, Principal Investigator — University Hospital of Aarhus
Locations (1):
- University Hospital of Aarhus, Norrebrogade, Aarhus, Denmark

REFERENCES:
- [Derived] Hjelholt AJ, Lee KY, Arlien-Soborg MC, Pedersen SB, Kopchick JJ, Puri V, Jessen N, Jorgensen JOL. Temporal patterns of lipolytic regulators in adipose tissue after acute growth hormone exposure in human subjects: A randomized controlled crossover trial. Mol Metab. 2019 Nov;29:65-75. doi: 10.1016/j.molmet.2019.08.013. Epub 2019 Aug 20. PMID 31668393
- [Derived] Nellemann B, Vendelbo MH, Nielsen TS, Bak AM, Hogild M, Pedersen SB, Bienso RS, Pilegaard H, Moller N, Jessen N, Jorgensen JO. Growth hormone-induced insulin resistance in human subjects involves reduced pyruvate dehydrogenase activity. Acta Physiol (Oxf). 2014 Feb;210(2):392-402. doi: 10.1111/apha.12183. Epub 2013 Nov 22. PMID 24148194